CLINICAL TRIAL: NCT03122158
Title: The Effect and Reliability of Escitalopram in the Treatment of Adolescents With Major Depressive Disorder or Anxiety Disorders
Brief Title: Escitalopram in the Treatment of Adolescents With Major Depressive Disorder or Anxiety Disorders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erzurum Regional Training & Research Hospital (Other Government)
Responsible Party: Principal Investigator, Muharrem Burak Baytunca, Child Psychiatry Consultant, MD, Erzurum Regional Training & Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ErzurumRTRH
Record Dates: First submitted 2017-04-08; First posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder; Anxiety Disorders
Keywords: major depressive disorder; anxiety disorders; adolescent; child
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders | interventions — Escitalopram

STUDY DESIGN:
Intervention Model Description: Adolescents with major depressive disorder or anxiety disorders will be recruited into 2 different diagnostic groups. Each group will include 30 participants. The total scores of the relevant assessment tools (Clinical Global Impression scale, Hamilton Rating Scale for Depression and Anxiety Disorders) at the starting point, 2nd and 6th month of the treatment will be compared.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Major depressive disorder (Active Comparator): In this group, adolescents with major depressive disorder will be recruited. It was planned to include 30 participants.Escitalopram treatment will be given to those with Major Depressive Disorder with a starting dose of 2.5 mg day. The treatment dose will be gradually increased up to 20 mg day (if necessary) and the maximal treatment dose was determined as 30 mg day in each group.
  Interventions: Drug: Escitalopram
- Anxiety disorders (Active Comparator): In this group, adolescents with anxiety disorders will be recruited. It was planned to include 30 participants. Additionally, the specification of which anxiety disorders are assigned to the participants will also be provided. Escitalopram treatment will be given to participants with anxiety disorders with a starting dose of 2.5 mg day. The treatment dose will be gradually increased up to 20 mg day (if necessary) and the maximal treatment dose was determined as 30 mg day in each group.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram treatment will be given to the arms with a starting dose of 2.5 mg day. The treatment dose will be gradually increased up to 20 mg day (if necessary) and the maximal treatment dose was determined as 30 mg day in each group.
  Other Names: Lexapro

SUMMARY:
Escitalopram has been approved by FDA in the treatment of adolescents with major depressive disorder since March 2009. To date, there are only 3 clinical trials assessing the effect and validity of escitalopram on major depressive disorder, which of them has resulted in inconsistent findings. In the present study, the authors aimed to assess the effect and validity of this drug in the treatment of adolescents with major depressive disorder and or anxiety disorders.

DETAILED DESCRIPTION:
Escitalopram has been approved by FDA in the treatment of adolescents with major depressive disorder since March 2009. Although Wagner and colleagues reported that escitalopram has a tendency toward positive findings for the treatment of pediatric patients with major depressive disorder in their study it was found that this effect has not reached a statistical significance. Noteworthy the authors reported statistical significance for escitalopram when they only included adolescent subgroup into further analysis. However, there are also clinical trials in the literature reporting the effectiveness of escitalopram on adolescence major depressive disorder (Emslie, Findling). It was indicated that no serious adverse effect of escitalopram was reported in these studies comparing escitalopram with placebo. In this study the authors aimed to investigate the effect and reliability of the drug in the treatment of adolescents with major depressive disorder and/or anxiety disorders. Additionally, cognitive behavioral therapy and SSRIs are indicated for the first-line treatment of anxiety disorders. The authors included escitalopram for the treatment of pediatric anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* drug-naive
* being in the age range of 12-18
* lack of any psychiatric comorbidity, except for ADHD-like problems during the illness
* IQ level> 80
* lack of history of any major medical disease, substance abuse

Exclusion Criteria:

* inappropriate age
* history of drug abuse, major medical disease
* mental retardation
* any psychotropic drug use
* hospitalization required for suicidal ideation/behavior

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-08 (Actual); Primary Completion 2018-09-15 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression Scale (CGI) | will be assessed in the 1st, 2nd and 6th month of the treatment.
  The authors will compare 3-time points of the treatment in the study. The first assessment point will be the starting point of the study and the other ones are 2nd and 6th months of the treatment course. Total scores of the CGI scale of the 3-time points will be recorded. Change in the scores of the starting point and 2nd month of the treatment will be compared. A decrease in the CGI score at the 2nd month of the treatment with a percentage of 50% or above will be considered as positive treatment response. The CGI score at the 6th month of the study with a result of 2 points or below will be accepted as remission.
The Hamilton Rating Scale for Depression | will be assessed in the 1st, 2nd and 6th month of the treatment in major depressive disorder arm.
  The authors will compare 3-time points of the treatment in the study. The first assessment point will be the starting point of the study and the other ones are 2nd and 6th months of the treatment course. Total scores of the Hamilton Depression scale of the 3-time points will be recorded. Change in the scores of the starting point and 2nd month of the treatment will be compared. A decrease in the Hamilton Depression scale score at the 2nd month of the treatment with a percentage of 50% or above will be considered as positive treatment response. Any scores on the Hamilton Depression scale below 8 points at the 6th month of treatment course will be accepted as remission.
The Hamilton Anxiety Rating Scale | will be assessed in the 1st, 2nd and 6th month of the treatment in anxiety disorders arm.
  The authors will compare 3-time points of the treatment in the study. The first assessment point will be the starting point of the study and the other ones are 2nd and 6th months of the treatment course. Total scores of the Hamilton Anxiety scale of the 3-time points will be recorded. Change in the scores of the starting point and 2nd month of the treatment will be compared. A decrease in the Hamilton Anxiety score at the 2nd month of the treatment with a percentage of 50% or above will be considered as positive treatment response. Any scores on the Hamilton Anxiety scale below 15 points at the 6th month of treatment course will be accepted as remission.

CONTACTS AND LOCATIONS:
Overall Officials: Muharrem Burak Baytunca, Principal Investigator — Erzurum Regional Training & Research Hospital
Locations (1):
- ErzurumRTRH, Erzurum, Palandöken, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
clinical severity of the participants measured by psychiatric tools and mean drug dose will be shared during the course of the study

REFERENCES:
- [Background] Wagner KD, Robb AS, Findling RL, Jin J, Gutierrez MM, Heydorn WE. A randomized, placebo-controlled trial of citalopram for the treatment of major depression in children and adolescents. Am J Psychiatry. 2004 Jun;161(6):1079-83. doi: 10.1176/appi.ajp.161.6.1079. PMID 15169696
- [Background] Emslie GJ, Ventura D, Korotzer A, Tourkodimitris S. Escitalopram in the treatment of adolescent depression: a randomized placebo-controlled multisite trial. J Am Acad Child Adolesc Psychiatry. 2009 Jul;48(7):721-729. doi: 10.1097/CHI.0b013e3181a2b304. PMID 19465881
- [Background] Findling RL, Robb A, Bose A. Escitalopram in the treatment of adolescent depression: a randomized, double-blind, placebo-controlled extension trial. J Child Adolesc Psychopharmacol. 2013 Sep;23(7):468-80. doi: 10.1089/cap.2012.0023. PMID 24041408